CLINICAL TRIAL: NCT00507793
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Cyclosporine Reduction in de Novo Renal Allograft Recipients Receiving Sirolimus: a Dose Comparative Study
Brief Title: Study Evaluating the Efficacy and Safety of Cyclosporine Reduction in Kidney Transplant Recipients Receiving Sirolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E1-4351
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2007-07-27 (Estimated); Status verified 2007-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sirolimus; Cyclosporine

INTERVENTIONS:
Drug: Sirolimus
Drug: Cyclosporine

SUMMARY:
To evaluate the safety and efficacy of different doses of cyclosporine given concomitantly with a fixed dose of sirolimus in kidney transplant recipients.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of different doses of cyclosporine given concomitantly with a fixed dose of sirolimus in kidney transplant recipients. Cyclosporine blood levels, graft rejection rates and renal function will be assessed.

ELIGIBILITY:
Inclusion criteria

* At least 18 years of age
* End-stage renal disease in patients receiving a primary or secondary renal allograft from a cadaveric, living-unrelated, or living-related mismatched donor
* Patients with secondary kidney transplant must have maintained primary graft for at least 6 months

Exclusion criteria

* Antibody induction within one week of current transplantation
* Multiorgan transplants
* Patients at high-risk of rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2000-04; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
A dose response model using the average cyclosporine blood levels correlated to graft rejection rates and renal function will be used to compare efficacy and safety of different doses of cyclosporine.

SECONDARY OUTCOMES:
Safety evaluations will include physical exams, vital signs, CBC with differential, platelet count, blood chemistries, fasting lipid profiles, BUN or urea, serum creatinine, adverse event monitoring and calculated creatinine clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Muhlbacher F, Neumayer HH, del Castillo D, Stefoni S, Zygmunt AJ, Budde K; European Rapamune Cyclosporine Minimization Study Group. The efficacy and safety of cyclosporine reduction in de novo renal allograft patients receiving sirolimus and corticosteroids: results from an open-label comparative study. Transpl Int. 2014 Feb;27(2):176-86. doi: 10.1111/tri.12228. Epub 2013 Nov 25. PMID 24266855